CLINICAL TRIAL: NCT02442778
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy, Safety, and Tolerability of AVP-786 (Deuterated [d6]-Dextromethorphan Hydrobromide [d6-DM]/Quinidine Sulfate [Q]) for the Treatment of Agitation in Patients With Dementia of the Alzheimer's Type
Brief Title: Efficacy, Safety, and Tolerability of AVP-786 for the Treatment of Agitation in Participants With Dementia of the Alzheimer's Type
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-AVP-786-302
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Results first posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-08

CONDITIONS: Agitation in Participants With Dementia of the Alzheimer's Type

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants were administered AVP-786 matching placebo capsules, orally, twice daily (BID) for up to 12 weeks.
  Interventions: Drug: Placebo
- AVP-786-28 (Experimental): Participants were administered AVP-786-18 capsule, orally, once daily (QD) along with AVP-786 matching placebo capsule, orally, QD during Week 1 followed by AVP-786-18 capsules, orally, BID during Weeks 2, 3 and AVP-786-28 capsules, orally, BID during Weeks 4 to 12.
  Interventions: Drug: AVP-786-18; Drug: AVP-786-28
- AVP-786-42.63 (Experimental): Participants were administered AVP-786-28 capsules, orally, QD along with AVP-786 matching placebo capsule, orally, QD during Week 1 followed by AVP-786-28 capsules, orally, BID during Weeks 2, 3, and AVP-786-42.63 capsules, orally, BID during Weeks 4 to 12.
  Interventions: Drug: AVP-786-28; Drug: AVP-786-42.63

INTERVENTIONS:
Drug: AVP-786-18 — 18 mg of Deudextromethorphan hydrobromide (d6-DM) and 4.9 mg of Quinidine sulfate (Q)
  Arms: AVP-786-28
Drug: Placebo — Administered as capsules.
  Arms: Placebo
Drug: AVP-786-28 — 28 mg of d6-DM and 4.9 mg of Q
  Arms: AVP-786-28; AVP-786-42.63
Drug: AVP-786-42.63 — 42.63 mg of d6-DM and 4.9 mg of Q
  Arms: AVP-786-42.63

SUMMARY:
Participants with agitation secondary to dementia of the Alzheimer's type. The diagnosis of probable Alzheimer's disease (AD) will be based on the "2011 Diagnostic Guidelines for Alzheimer's Disease" issued by the National Institute on Aging (NIA)-Alzheimer's Association (AA) workgroups.

DETAILED DESCRIPTION:
Eligible participants for this study must have a diagnosis of probable AD and must have clinically meaningful agitation secondary to AD.

This is a multicenter, randomized, placebo-controlled study, consisting of 12 weeks of treatment.

Approximately 470 participants will be enrolled at approximately 75 centers in North America.

Study medication will be administered orally twice-daily from Day 1 through Week 12 (Day 85). Screening will occur within approximately 4 weeks prior to randomization. Following screening procedures for assessment of inclusion and exclusion criteria, eligible participants will be randomized into the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's Disease (AD) according to the 2011 National Institute on Aging-Alzheimer's Association (NIA-AA) working groups criteria
* The participant has clinically significant, moderate/severe agitation at the time of screening and for at least 2 weeks prior to randomization
* The diagnosis of agitation must meet the International Psychogeriatric Association (IPA) provisional definition of agitation
* Either out participants or residents of an assisted-living facility or a skilled nursing home
* Clinical Global Impression of Severity of Illness (CGIS) score assessing Agitation is >=4 (moderately ill) at screening and baseline
* Mini-Mental State Examination (MMSE) score is between 6 and 26 (inclusive) at screening and baseline
* Caregiver who is able and willing to comply with all required study procedures. In order to qualify as a reliable informant (i.e., caregiver) capable of assessing changes in participant's condition during the study, the individual must spend a minimum of 2 hours per day for 4 days per week with the participant.

Exclusion Criteria:

* Participant has dementia predominantly of non-Alzheimer's type (e.g., vascular dementia, frontotemporal dementia, Parkinson's disease, substance-induced dementia)
* Participants with co-existent clinically significant or unstable systemic diseases that could confound the interpretation of the safety results of the study (e.g., malignancy, poorly controlled diabetes, poorly controlled hypertension, unstable pulmonary, renal or hepatic disease, unstable ischemic cardiac disease, dilated cardiomyopathy, or unstable valvular heart disease)
* Participant with myasthenia gravis

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (83):
- United States (79):
  - Brain and Spine Center, Chandler, Arizona
  - Territory Neurology & Research Institute, Tucson, Arizona
  - Health Initiatives Research, Fayetteville, Arkansas
  - Behavioral Research Specialists, LLC, Glendale, California
  - Irvine Center for Clinical Research, Irvine, California
  - California Neurological Services, Panorama City, California
  - Havana Research Institute, Pasadena, California
  - Pacific Research Network, Inc, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Viking Clinical Research, Temecula, California
  - Denver Neurological Research, LLC, Denver, Colorado
  - JEM Research Institute, Atlantis, Florida
  - Clinical Research Of Brandon, LLC, Brandon, Florida
  - Meridien Research, Brooksville, Florida
  - Moonshine Research Center, Inc, Doral, Florida
  - Science Connections, LLC, Doral, Florida
  - Finlay Medical Research Corp, Greenacres City, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - New Life Medical Research Center, Inc., Hialeah, Florida
  - Reliable Clinical Research,LLC, Hialeah, Florida
  - Research in Miami, Inc, Hialeah, Florida
  - The Research Center, Inc, Hialeah, Florida
  - Maxblue Institute, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Alzheimer's Research and Treatment Center, Lake Worth, Florida
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - Project 4 Research, Miami, Florida
  - BioMed Research Institute, Miami, Florida
  - CCM Clinical Research Group, Miami, Florida
  - DADE Research Center, LLC, Miami, Florida
  - AMB Research Center, Inc., Miami, Florida
  - United Health Research Corp, Miami, Florida
  - Advance Medical Research Center, Miami, Florida
  - Coral Research Clinic Corp, Miami, Florida
  - P&S Reasearch, Miami, Florida
  - The Neurology Research Group, LLC, Miami, Florida
  - Kendall Research Institute, Miami, Florida
  - Nuovida Research Center Corp., Miami, Florida
  - Collier Neurologic Specialists, LLC, Naples, Florida
  - Lazlo J. Mate, MD, PA, North Palm Beach, Florida
  - Compass Research, LLC, Orlando, Florida
  - IMIC Inc., Palmetto Bay, Florida
  - University of West Florida, Pensacola, Florida
  - Neurology Research Institute Palm Beach, LLC, West Palm Beach, Florida
  - Emory Brain Health Center, Atlanta, Georgia
  - Columbus Research & Wellness Institute, INC, Columbus, Georgia
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - Baptist Health Medical Group, Richmond, Kentucky
  - The Samuel & Alexia Bratton Memory Clinic, Easton, Maryland
  - Mir Neurology, Hagerstown, Maryland
  - Boston Center for Memory, Newton, Massachusetts
  - AMAC Research Institute, North Dartmouth, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - The NeuroCognitive Institute, Mount Arlington, New Jersey
  - Brooklyn Medical Institute, Brooklyn, New York
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - Eastside Comprehensive Medical Center, LLC, New York, New York
  - Burke Rehabilitation Hospital, White Plains, New York
  - Herbert Harris, MD, PhD, PA, Chapel Hill, North Carolina
  - ANI Neurology PLLC dba Alzheimer's Memory Center, Charlotte, North Carolina
  - Daystar Clinical Research Inc, Akron, Ohio
  - Valley Medical Research, Centerville, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Cleveland Clinic Lou Ruvo Center for Brain Health at Lakewood Hospital, Lakewood, Ohio
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - The Birches at Newton / Family Medical Associates, Levittown, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - RH Johnson VA Medical Center, Charleston, South Carolina
  - BG Neurology, Spartanburg, South Carolina
  - Texas Neurology, P.A., Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Texas Medical Research Associates, L.L.C., San Antonio, Texas
  - Pharmaceuticals Research Associates, Inc., Salt Lake City, Utah
  - Clinical Neuroscience Research Associates, Inc. dba The Memory Clinic, Bennington, Vermont
  - Veteran Affairs Medical Center, Salem Virginia, Salem, Virginia
  - IPC Research, Waukesha, Wisconsin
- Canada (4):
  - Dr. Alexander McIntyre Inc., Calgary, Alberta
  - The Medical Art Health Research Group, Kelowna, Bristish Columbia
  - The Medical Art Health Research Group, Penticton, Bristish Columbia
  - The Medical Art Health Research Group, West Vancouver, Bristish Columbia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researcher sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publica data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/O
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 83 investigative sites in North America from 11 November 2015 to 09 September 2019.
Pre-assignment Details: A total of 925 participants were screened of which 522 participants were enrolled and 521 participants were randomized to receive placebo or AVP-786-28 or AVP-786-42.63.
Groups:
- AVP-786-42.63: Participants were administered AVP-786-28 capsule, orally, QD along with AVP-786 matching placebo capsule, orally, QD during Week 1 followed by AVP-786-28 capsules, orally, BID during Weeks 2, 3 and AVP-786-42.63 capsules, orally, BID during Weeks 4 to 12.
Period: Overall Study
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Started | 210 | 151 | 161
Safety Population (Safety Population included all participants who received at least one dose of study medication. Participants were included in the treatment group based on the actual treatment received.) | 210 | 151 | 160
Modified Intent-to-Treat (mITT) Population (mITT Population included all randomized participants who had at least one post-baseline efficacy assessment. Participants were included in the treatment group to which they were randomized regardless of treatment received) | 210 | 150 | 159
Completed | 192 | 121 | 146
Not Completed | 18 | 30 | 15
Not completed — Adverse Event | 2 | 6 | 6
Not completed — Death | 0 | 2 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Non-compliance with study drug | 2 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Protocol Deviation | 3 | 0 | 1
Not completed — Study participant withdrawal by parent or guardian | 3 | 12 | 2
Not completed — Withdrawal by Subject | 4 | 4 | 3
Not completed — Reason not specified | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized Population included all the participants who were randomized in the study.
Groups:
- Placebo: Participants were administered AVP-786 matching placebo capsules, orally, BID for up to 12 weeks.
- AVP-786-28: Participants were administered AVP-786-18 capsule, orally, QD along with AVP-786 matching placebo capsule, orally, QD during Week 1 followed by AVP-786-18 capsules, orally, BID during Weeks 2, 3 and AVP-786-28 capsules, orally, BID during Weeks 4 to 12.
- Total: Total of all reporting groups
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63 | Total
Number analyzed (Participants) | 210 | 151 | 161 | 522
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.7 (8.1) | 74.6 (7.9) | 74.8 (7.3) | 75.5 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 84 | 96 | 297
  Male | 93 | 67 | 65 | 225
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 196 | 129 | 155 | 480
  Race: Black or African American | 13 | 14 | 6 | 33
  Race: Asian | 0 | 2 | 0 | 2
  Race: American Indian or Alaska Native | 1 | 0 | 0 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Race: Other | 0 | 5 | 0 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 128 | 78 | 113 | 319
  Ethnicity: Not Hispanic or Latino | 82 | 73 | 48 | 203

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Cohen-Mansfield Agitation Inventory (CMAI) Composite Score
Description: The CMAI was used to assess the frequency of manifestations of agitated behaviors in elderly participants. It consists of 29 agitated items rated on a 7-point scale of frequency: 1, never; 2, less than once a week; 3, once or twice a week; 4, several times a week; 5, once or twice a day; 6, several times a day; 7, several times an hour. The CMAI total score ranges from 29 to 203. Higher scores indicate worsening of the condition. Negative change from baseline indicates improvement. Mixed Model Repeated Measures (MMRM) was used for the analysis.
Time Frame: Baseline, Week 12
Population: mITT Population included all randomized participants who had at least one post-baseline efficacy assessment. Participants were included in the treatment group to which they were randomized regardless of treatment received. Number analysed signifies the number of participants with available data for analysis at a specific timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 210 | 150 | 159
score on a scale
  Baseline | 73.7 (21.13) | 68.8 (19.39) | 71.3 (20.87)
  Change from Baseline at Week 12: number analyzed (Participants) | 188 | 120 | 141
  Change from Baseline at Week 12 | -16.2 (16.97) | -12.7 (16.21) | -17.0 (16.12)
Statistical Analysis 1: Comparison: Placebo vs AVP-786-28; Test type: Superiority; p = 0.789, MMRM — MMRM included fixed effect treatment,visit,treatment-by-visit,baseline,baseline-by-visit,baseline Neuropsychiatric Inventory Agitation/Aggression(NPI AA)(≤6 vs. >6),falls risk assessment,baseline concomitant use of antipsychotic medications,cohorts; Least Squares (LS) Mean Difference = 0.4, 95% CI 2-sided [-2.7 to 3.5]
Statistical Analysis 2: Comparison: Placebo vs AVP-786-42.63; Test type: Superiority; p = 0.200, MMRM — MMRM included fixed effect treatment, visit, treatment-by-visit, baseline, baseline-by-visit, baseline NPI AA (≤ 6 vs. > 6), risk assessment for falls, baseline concomitant use of antipsychotic medications and cohorts; LS Mean Difference = -2.0, 95% CI 2-sided [-5.0 to 1.0]

2. Secondary Outcome: Relative Change From Baseline to Week 12 in the Modified Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (mADCS-CGIC)-Agitation Score
Description: The mADCS-CGIC-Agitation is a modified version of the ADCS-CGIC containing additional questions related to agitation and an assessment of the Clinician's Impression of Change focused specifically on agitation. Participants are asked to rate their impression of change as: 1=Marked Improvement; 2=Moderate Improvement; 3=Minimal Improvement; 4=No Change; 5=Minimal Worsening; 6=Moderate Worsening; 7=Marked Worsening. Higher scores indicate worsening of agitation and positive change from baseline indicates worsening. MMRM was used for the analysis.
Time Frame: Baseline, Week 12
Population: mITT Population included all randomized participants who had at least one post-baseline efficacy assessment. Participants were included in the treatment group to which they were randomized regardless of treatment received. Overall number of participants analysed signifies the number of participants with available data for analysis at specific timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 190 | 118 | 141
score on a scale | 2.9 (1.18) | 3.1 (1.23) | 2.8 (1.20)
Statistical Analysis 1: Comparison: Placebo vs AVP-786-28; Test type: Superiority; p = 0.484, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.2 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs AVP-786-42.63; Test type: Superiority; p = 0.704, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.2]

3. Secondary Outcome: Change From Baseline to Week 12 in the Neuropsychiatric Inventory (NPI) Agitation/Aggression Domain Score
Description: The NPI is a retrospective caregiver-informant interview covering 12 neuropsychiatric symptom domains. The Agitation/Aggression domain is designed to collect information on the behavioral aspects of agitation/aggression in participants with probable AD and clinically meaningful agitation secondary to AD. Each NPI domain is rated by the caregiver for symptom frequency and severity. Symptom frequency is rated as:1, occasionally; 2, often; 3, frequently; 4, very frequently. Symptom severity is rated as: 1, mild; 2, moderate; 3, severe. The total domain score is calculated as the frequency score multiplied by the severity score and thus ranges from 1 to 12. Higher scores indicate worsening symptoms. Negative change from baseline indicates improvement in symptoms. MMRM was used for the analysis.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 192 | 123 | 148
score on a scale | -2.5 (3.17) | -2.3 (3.32) | -3.2 (3.32)
Statistical Analysis 1: Comparison: Placebo vs AVP-786-28; Test type: Superiority; p = 0.416, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.9 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs AVP-786-42.63; Test type: Superiority; p = 0.066, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.6, 95% CI 2-sided [-1.3 to 0.0]

4. Secondary Outcome: Change From Baseline to Week 12 in the NPI Agitation/Aggression Caregiver Distress Score
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate caregiver distress. Each NPI domain is rated by the caregiver for symptom frequency and severity. Symptom frequency is rated as:1, occasionally; 2, often; 3, frequently; 4, very frequently. Symptom severity is rated as:1, mild; 2, moderate; 3, marked severe. The total caregiver distress score is calculated as the frequency score multiplied by the severity score and thus ranges from 1 to 12 with a higher score indicating worsening of symptoms. Negative change from baseline indicates improvement in symptoms. MMRM was used for the analysis.
Time Frame: Baseline, Week 12
Population: mITT Population included all randomized participants who had at least one post-baseline efficacy assessment. Participants were included in the treatment group to which they were randomized regardless of treatment received. Overall number of participants analysed signifies the number of participants with available data for analysis at a specific timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 189 | 121 | 144
score on a scale | -0.8 (1.44) | -0.8 (1.61) | -0.8 (1.47)
Statistical Analysis 1: Comparison: Placebo vs AVP-786-28; Test type: Superiority; p = 0.249, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.1]
Statistical Analysis 2: Comparison: Placebo vs AVP-786-42.63; Test type: Superiority; p = 0.199, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.1]

5. Secondary Outcome: Change From Baseline to Week 12 in the NPI Aberrant Motor Behavior Domain Score
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate aberrant motor behavior. Each NPI domain is rated by the caregiver for symptom frequency and severity. Symptom frequency is rated as: 1, occasionally; 2, often; 3, frequently; 4, very frequently. Symptom severity is rated as: 1, mild; 2, moderate; 3, marked severe. The total domain score is calculated as the frequency score multiplied by the severity score and thus ranges from 1 to 12 with a higher score indicating worsening of symptoms. Negative change from baseline indicates improvement in symptoms. MMRM was used for the analysis.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 192 | 123 | 148
score on a scale | -1.2 (3.75) | -1.2 (3.60) | -1.8 (3.57)
Statistical Analysis 1: Comparison: Placebo vs AVP-786-28; Test type: Superiority; p = 0.975, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.7 to 0.7]
Statistical Analysis 2: Comparison: Placebo vs AVP-786-42.63; Test type: Superiority; p = 0.334, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.3, 95% CI 2-sided [-1.0 to 0.3]

6. Secondary Outcome: Change From Baseline to Week 12 in the Zarit Burden Interview (ZBI) Score
Description: The ZBI is a 22-item scale used to assess the impact of a participants' disabilities on the caregiver's life. It is designed to reflect the burden experienced by caregivers of dementia participants and can either be completed by the caregiver or administered as an interview. Each item of the scale is rated to reflect the burden using the 5-point scale: 0=Never; 1=Rarely; 2=Sometimes; 3=Quite Frequently; 4=Nearly Always. The ZBI is scored by summing the responses of the individual questions and ranges from 0 to 88. Higher scores indicate greater caregiver distress. Negative change from baseline indicates less distress. MMRM was used for the analysis.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 190 | 118 | 141
score on a scale | -1.77 (9.275) | -1.03 (12.195) | -0.23 (11.769)
Statistical Analysis 1: Comparison: Placebo vs AVP-786-28; Test type: Superiority; p = 0.934, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.1, 95% CI 2-sided [-2.4 to 2.2]
Statistical Analysis 2: Comparison: Placebo vs AVP-786-42.63; Test type: Superiority; p = 0.342, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 1.1, 95% CI 2-sided [-1.2 to 3.4]

7. Secondary Outcome: Change From Baseline to Week 12 in the NPI Irritability/Lability Domain Score
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains, including the irritability/lability domain score. Each NPI domain is rated by the caregiver for symptom frequency and severity. Symptom frequency is rated as:1, occasionally; 2, often; 3, frequently; 4, very frequently. Symptom severity is rated as:1, mild; 2, moderate; 3, severe. The total domain score is calculated as the frequency score multiplied by the severity score and thus ranges from 1 to 12. Higher scores indicate worsening of the symptoms. Negative change from baseline indicates improvement in symptoms. MMRM was used for the analysis.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 192 | 123 | 148
score on a scale | -1.8 (3.50) | -1.2 (3.55) | -2.2 (3.29)
Statistical Analysis 1: Comparison: Placebo vs AVP-786-28; Test type: Superiority; p = 0.888, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.0, 95% CI 2-sided [-0.7 to 0.6]
Statistical Analysis 2: Comparison: Placebo vs AVP-786-42.63; Test type: Superiority; p = 0.019, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.7, 95% CI 2-sided [-1.3 to -0.1]

8. Secondary Outcome: Change From Baseline to Week 12 in the NPI Total Score
Description: NPI evaluates both frequency and severity of 12 neuropsychiatric disturbances including delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, night time behaviors, as well as appetite/eating. Total domain score= frequency x severity and thus ranges from 1 to 12. NPI domain is rated by caregiver for symptom frequency and severity. Frequency is rated as:1=occasionally, 2=often, 3= frequently, and 4=very frequently. Severity is rated as:1=mild,2=moderate,3=severe. Frequency and severity rating scales has defined anchor points to enhance reliability of caregiver responses. Caregiver distress is rated for each positive neuropsychiatric symptom using following anchored scores. It is rated as 0=not at all,1=minimal,2=mild,3=moderate,4=severe,5=very severe. Individual Item scores are added to yield a possible total score of 0 to 144. MMRM was used for the analysis.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 192 | 123 | 148
score on a scale | -12.3 (17.06) | -9.5 (18.41) | -16.9 (18.05)
Statistical Analysis 1: Comparison: Placebo vs AVP-786-28; Test type: Superiority; p = 0.756, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.6, 95% CI 2-sided [-2.9 to 4.0]
Statistical Analysis 2: Comparison: Placebo vs AVP-786-42.63; Test type: Superiority; p = 0.038, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -3.6, 95% CI 2-sided [-7.0 to -0.2]

9. Secondary Outcome: Change From Baseline to Week 12 in the Clinical Global Impression of Severity of Illness (CGIS)-Agitation Domain Score
Description: The CGIS-Agitation is an observer-rated scale that measures illness severity. The CGIS-Agitation is a 7-point (1-7) scale (1=normal, not at all ill participants; 7=among the most extremely ill participants) and is assessed for severity of agitation. A value of 0 is given to participants who are not assessed. Higher scores indicate poor health of participants. MMRM was used for the analysis.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 190 | 118 | 141
score on a scale | -0.7 (0.85) | -0.7 (0.92) | -0.8 (0.93)
Statistical Analysis 1: Comparison: Placebo vs AVP-786-28; Test type: Superiority; p = 0.468, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1]
Statistical Analysis 2: Comparison: Placebo vs AVP-786-42.63; Test type: Superiority; p = 0.158, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1]

10. Secondary Outcome: Change From Baseline to Week 12 in the Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) Overall Rating
Description: The ADCS-CGIC rating scale provides a reliable means to assess change from a Baseline level of global function within the time frame of the trial. ADCS-CGIC-Overall focuses on the clinician's observations of change in the participant's cognitive, functional, and behavioral performance. The ADCS-CGIC-Overall responses (1-7) are rated as: 1 = marked improvement, 2 = moderate improvement, 3 = minimal improvement, 4 = no change, 5 = minimal worsening, 6 = moderate worsening, or 7 = marked worsening. MMRM was used for the analysis.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 188 | 118 | 141
score on a scale | 3.2 (1.20) | 3.4 (1.31) | 3.1 (1.23)
Statistical Analysis 1: Comparison: Placebo vs AVP-786-28; Test type: Superiority; p = 0.400, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.2 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs AVP-786-42.63; Test type: Superiority; p = 0.566, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.2]

11. Secondary Outcome: Change From Baseline to Week 12 in the Patient Global Impression of Change (PGIC) Score
Description: The PGIC is a 7-point (1-7) scale used to assess treatment response: 1 = very much improved, = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, or 7 = very much worse. Higher scores indicate less response to treatment. MMRM was used for the analysis.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 191 | 118 | 141
score on a scale | 3.1 (1.01) | 3.1 (1.07) | 2.9 (1.05)
Statistical Analysis 1: Comparison: Placebo vs AVP-786-28; Test type: Superiority; p = 0.751, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs AVP-786-42.63; Test type: Superiority; p = 0.320, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1]

12. Secondary Outcome: Change From Baseline to Week 12 in the Dementia Quality of Life (DEMQOL) Score
Description: The DEMQOL scale is used to evaluate health-related QOL in participants with dementia and their caregivers. There are 2 versions of the DEMQOL: a 28-item version (rated by the participant); and a 31-item version (DEMQOL-proxy, rated by the caregiver). Both versions are recommended for evaluating participants (and their caregivers) with mild to moderate dementia. The DEMQOL total score ranges from 28 to 112. The DEMQOL-proxy is used for participants with severe dementia; the total score ranges from 31 to 124. For both versions, higher scores indicate greater QOL. MMRM was used for the analysis.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 153 | 96 | 117
score on a scale | 2.9 (11.10) | 3.8 (8.10) | 3.2 (8.74)
Statistical Analysis 1: Comparison: Placebo vs AVP-786-28; Test type: Superiority; p = 0.782, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.3, 95% CI 2-sided [-1.8 to 2.4]
Statistical Analysis 2: Comparison: Placebo vs AVP-786-42.63; Test type: Superiority; p = 0.991, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.0, 95% CI 2-sided [-2.1 to 2.0]

13. Secondary Outcome: Change From Baseline in the Cornell Scale for Depression in Dementia (CSDD) Score
Description: The CSDD scale is used to assess signs/symptoms of major depression in participants with dementia. CSDD has 19 items, and each item is rated for severity on the following scale of 0 to 2 (0 =absent, 1= mild/intermittent 2=severe). CSDD score is calculated by summing non-missing scores from each item score. The scale ranges from 0 (no depression) to 38 (maximum depression). Scores above 10 indicate a probable major depression, above 18 indicate a definite major depression, and below 6 as a rule are associated with the absence of significant depressive symptoms. Higher score indicated maximum depression. MMRM was used for the analysis.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 189 | 118 | 141
score on a scale | -1.1 (2.84) | -0.5 (2.90) | -1.5 (2.57)
Statistical Analysis 1: Comparison: Placebo vs AVP-786-28; Test type: Superiority; p = 0.038, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.6, 95% CI 2-sided [0.0 to 1.2]
Statistical Analysis 2: Comparison: Placebo vs AVP-786-42.63; Test type: Superiority; p = 0.911, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.0, 95% CI 2-sided [-0.6 to 0.5]

14. Secondary Outcome: Number of Participants With the Change From Baseline in the General Medical Health Rating (GMHR) Score at Week 12
Description: The GMHR is a global clinical rating for medical health, designed to quantify in a single number (1 to 4) the severity of general comorbidity in a participant with dementia. The ratings are: 1 = poor; 2 = fair; 3 = good; 4 = excellent to very good. MMRM was used for the analysis.
Time Frame: Week 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 210 | 150 | 158
Participants
  Fair to Excellent to Very Good | 6 | 6 | 3
  Poor to Excellent to Very Good | 22 | 7 | 10
  Good to Good | 17 | 9 | 10
  Fair to Good | 80 | 65 | 65
  Poor to Good | 6 | 6 | 4
  Missing to Good | 1 | 0 | 0
  Good to Fair | 53 | 31 | 43
  Fair to Fair | 11 | 6 | 11
  Poor to Fair | 0 | 3 | 1
  Fair to Poor | 1 | 0 | 0
  Good to Missing | 5 | 4 | 7
  Fair to Missing | 7 | 9 | 4
  Poor to Missing | 1 | 4 | 0

15. Secondary Outcome: Change From Baseline to Week 12 in the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) Score
Description: The ADAS is designed to evaluate the cognitive and non-cognitive behavioral dysfunction characteristics of participants with AD. The cognitive subscale (ADAS-cog) consists of 11 subsets related to memory, praxis, and language. ADAS-cog scores range from 0 to 70. Higher scores indicate greater cognitive impairment. Negative change from baseline indicates less cognitive impairment. MMRM method was used for analysis.
Time Frame: Baseline, Week 12
Population: mITT Population included all randomized participants who had at least one post-baseline efficacy assessment. Participants were included in the treatment group to which they were randomized regardless of treatment received. Overall number analysed signifies the number of participants with available data for analysis at specific timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 143 | 91 | 97
score on a scale | -2.0 (5.67) | -1.0 (7.36) | -1.5 (6.38)
Statistical Analysis 1: Comparison: Placebo vs AVP-786-28; Test type: Superiority; p = 0.236, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 1.0, 95% CI 2-sided [-0.6 to 2.6]
Statistical Analysis 2: Comparison: Placebo vs AVP-786-42.63; Test type: Superiority; p = 0.684, MMRM — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.3, 95% CI 2-sided [-1.3 to 1.9]

16. Secondary Outcome: Resource Utilization in Dementia (RUD) Score: Number of Hours Per Day the Caregiver Spent Assisting the Participant
Description: The RUD evaluates dementia participants' utilization of formal and informal healthcare resources, including hospitalizations and doctor visits, living assistance, and time spent by nonprofessional caregivers. Information on hours per day the caregiver spent assisting participant were reported in this outcome measure, using the following questions:
  Q1= On a typical care day during the last 30 days, how much time per day did you assist the participant with tasks such as toilet visits, eating, dressing, grooming, walking and bathing? Q2= On a typical care day during the last 30 days, how much time per day did you assist the participant with tasks such as shopping, food preparation, housekeeping, laundry, transportation, taking medication and managing financial matters? Q3= On a typical care day during the last 30 days, how much time per day did you spend supervising (that is, preventing dangerous events) the participant?
Time Frame: Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 210 | 150 | 159
hours
  Q1: number analyzed (Participants) | 173 | 111 | 136
  Q1 | 3.0 [0 to 24] | 3.0 [0 to 18] | 3.0 [0 to 24]
  Q2: number analyzed (Participants) | 173 | 111 | 136
  Q2 | 4.5 [0 to 24] | 5.0 [0 to 24] | 5.0 [0 to 24]
  Q3: number analyzed (Participants) | 173 | 111 | 136
  Q3 | 5.0 [0 to 24] | 4.0 [0 to 24] | 6.0 [0 to 24]

17. Secondary Outcome: Resource Utilization in Dementia (RUD) Score: Number of Days the Caregiver Spent Assisting the Participant
Description: The RUD evaluates dementia participants' utilization of formal and informal healthcare resources, including hospitalizations, doctor visits, living assistance, and time spent by nonprofessional caregivers. Information on days the caregiver spent assisting participant were reported in this outcome measure, using the following questions:
  Q1= During the last 30 days, how many days did you spend providing these (toilet visits, eating, dressing, grooming, walking and bathing) services to the participant? Q2= During the last 30 days, how many days did you spend providing these (shopping, food preparation, housekeeping, laundry, transportation, taking medication and managing financial matters) services to the participant? Q3= During the last 30 days, how many days did you spend providing these services (supervising) to the participant?
Time Frame: Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 210 | 150 | 159
days
  Q1: number analyzed (Participants) | 173 | 111 | 136
  Q1 | 30.0 [0 to 30] | 30.0 [0 to 30] | 30.0 [0 to 30]
  Q2: number analyzed (Participants) | 173 | 111 | 136
  Q2 | 30.0 [0 to 30] | 30.0 [0 to 30] | 30.0 [0 to 30]
  Q3: number analyzed (Participants) | 173 | 111 | 136
  Q3 | 30.0 [0 to 30] | 30.0 [0 to 30] | 30.0 [0 to 30]

18. Secondary Outcome: Resource Utilization in Dementia (RUD) Score: Number of Visits to Hospital, Emergency, and Healthcare Professional
Description: The RUD evaluates dementia participants' utilization of formal and informal healthcare resources, including hospitalizations, doctor visits, living assistance, and time spent by nonprofessional caregivers. Information on the number of hospital visits, emergency visits and visits to healthcare professional were reported in this outcome measure using the following questions:
  Q1= During the last 30 days, how many times did the participant receive care in a hospital emergency room (for less than 24 hours)? Q2= During the last 30 days, how many times did the caregiver receive care in a hospital emergency room (for less than 24 hours)? Q3= During the last 30 days total number of visits by participant to a health care professional? Q4= During the last 30 days, how many times (number of visits for each) the participant visited any other health care professional?
Time Frame: Week 12
Population: mITT Population included all randomized participants who had at least one post-baseline efficacy assessment. Participants were included in the treatment group to which they were randomized regardless of treatment received. Number analysed signifies the number of participants with available data for analysis at specific timepoint.
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
Number analyzed (Participants) | 210 | 150 | 159
Number of visits
  Q1: number analyzed (Participants) | 4 | 3 | 3
  Q1 | 1.0 (0.0) | 1.3 (0.58) | 1.3 (0.58)
  Q2: number analyzed (Participants) | 1 | 0 | 2
  Q2 | 1.0 (NA) — SD cannot be calculated for 1 participant. |  | 1.0 (0.00)
  Q3: number analyzed (Participants) | 173 | 109 | 130
  Q3 | 2.7 (1.35) | 2.5 (1.28) | 2.6 (1.45)
  Q4: number analyzed (Participants) | 167 | 101 | 126
  Q4 | 2.2 (0.88) | 2.1 (0.51) | 2.0 (0.59)

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days after the last dose of study drug (up to 16 weeks)
Description: All-cause mortality: All Randomized Population included all the participants who were randomized in the study.
  Adverse events: Safety Population included all participants who received at least one dose of study medication. Participants were included in the treatment group based on the actual treatment received.
Arm/Group | Placebo | AVP-786-28 | AVP-786-42.63
All-Cause Mortality (participants affected / at risk) | 0/210 | 3/151 | 0/161
Serious Adverse Events (participants affected / at risk) | 10/210 | 15/151 | 8/160
Other Adverse Events (participants affected / at risk) | 40/210 | 31/151 | 30/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=210) | AVP-786-28 (N=151) | AVP-786-42.63 (N=160)
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic insufficiency (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Administration site joint infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0
Influenza A virus test positive (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 3 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=210) | AVP-786-28 (N=151) | AVP-786-42.63 (N=160)
Diarrhoea (Gastrointestinal disorders) | 14 | 5 | 5
Urinary tract infection (Infections and infestations) | 11 | 10 | 3
Fall (Injury, poisoning and procedural complications) | 8 | 15 | 10
Somnolence (Nervous system disorders) | 2 | 4 | 11
Agitation (Psychiatric disorders) | 12 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT02442778/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT02442778/SAP_001.pdf